CLINICAL TRIAL: NCT01169636
Title: Phase I Study of Panobinostat Plus ICE Chemotherapy Followed by a Randomized Phase-II Study of ICE Compared With Panobinostat Plus ICE for Patients With Relapsed and Refractory Classical Hodgkin Lymphoma
Brief Title: Panobinostat Plus Ifosfamide, Carboplatin, and Etoposide (ICE) Compared With ICE For Relapsed Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0065; NCI-2012-01779 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Hodgkin's Lymphoma
Keywords: Chemotherapy; Panobinostat; Ifosfamide; Mesna; Etoposide; Carboplatin; Pegfilgrastim; ICE
MeSH Terms: conditions — Hodgkin Disease | interventions — Panobinostat; Ifosfamide; Mesna; Carboplatin; Etoposide; pegfilgrastim; pegylated granulocyte colony-stimulating factor, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Panobinostat MTD + ICE (Experimental): Phase 1: Escalating Panobinostat dose with routine ICE Chemotherapy
  Interventions: Drug: Panobinostat; Drug: Ifosfamide; Drug: Mesna; Drug: Carboplatin; Drug: Etoposide
- ICE Chemotherapy (Experimental): Phase 2: Routine ICE Chemotherapy (Ifosfamide, Carboplatin, + Etoposide)
  Interventions: Drug: Ifosfamide; Drug: Mesna; Drug: Carboplatin; Drug: Etoposide; Drug: Pegfilgrastim
- Panobinostat + ICE (Experimental): Phase 2: Panobinostat with ICE Chemotherapy
  Interventions: Drug: Panobinostat; Drug: Ifosfamide; Drug: Mesna; Drug: Carboplatin; Drug: Etoposide; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Panobinostat — Starting Day -6 of Cycle 1, 20 mg orally on Monday, Wednesday, and Friday during Cycles 1 and 2 (Days -6, -4, and -2 of Cycle 1 and Days 1, 3, 5, 8, 10, and 12 of Cycles 1 and 2); MTD found in Phase 1 used for same schedule in Phase 2.
  Other Names: LBH589B
  Arms: Panobinostat + ICE; Panobinostat MTD + ICE
Drug: Ifosfamide — Day 1 of Cycles 1-3, 5 grams/m2 by vein over 24 hours.
  Other Names: Ifex
Drug: Mesna — On Day 1 of Cycles 1-3, 2 grams/m2 by vein over 12 hours.
  Other Names: Mesnex
Drug: Carboplatin — On Day 1 of Cycles 1-3, Standard Dose (Target area under curve (AUC) = 5mg/ml/min) by vein over 1 hour.
  Other Names: Paraplatin
Drug: Etoposide — On Days 1-3 of Cycles 1-3, 100 mg/m2 by vein over 2 hours.
  Other Names: VePesid
Drug: Pegfilgrastim — Beginning Day 4 of Cycles 1-3, 6 mg under the skin.
  Other Names: Neulasta; PEG-G-CSF
  Arms: ICE Chemotherapy; Panobinostat + ICE

SUMMARY:
Objectives:

Primary objective:

* Phase-I: To determine the maximal tolerated dose (MTD) of panobinostat (LBH589) + Ifosfamide + Mesna, Carboplatin and Etoposide (ICE) combination
* Randomized Phase-II: To estimate the complete response (CR) rate in patients with relapsed and refractory classical Hodgkins Lymphoma (HL) receiving ICE versus PANOBINOSTAT plus ICE therapy

Secondary Objectives:

* To assess the safety and tolerability of the novel combination of PANOBINOSTAT (LBH589) plus ICE versus ICE in patients with relapsed and refractory HL
* To estimate the overall response rate (CR + partial response PR)
* To estimate the success rate of stem cell collection in patients eligible for stem cell transplant
* To estimate the percentage of patients who subsequently undergo autologous stem cell transplantation (ASCT)
* To estimate the event free survival (EFS) at 1 year after randomization
* To determine pretreatment expression level of histone deacetylases (HDAC1), HDAC2, and pSTAT3 and Signal transducer and activator of transcription protein (pSTAT6) by Immunohistochemistry (IHC) and correlate the results with treatment response

DETAILED DESCRIPTION:
Phase I:

The Study Drugs:

Panobinostat is designed to block the function of enzymes that are found inside cancer cells. These enzymes trigger cells to grow and multiply out of control. By blocking these enzymes, it may slow down the growth of or kill cancer cells.

Ifosfamide is designed to slow or stop the growth of cancer cells.

Carboplatin is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

Etoposide is designed to block cell growth.

Baseline Tests:

If you are found to be eligible to take part in this study, the following tests and procedures will be performed about 7 days before the first dose of the study drug:

* You will have a physical exam, including measurement of your height, weight, and vital signs (blood pressure and heart rate).
* You will have 1 electrocardiogram (ECG -- a test that measures the electrical activity of the heart).
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* Women who are able to become pregnant must have a negative blood (about 1 1/2 teaspoons) pregnancy test.

Study Groups:

You will be assigned to a dose level of panobinostat based on when you join this study. Up to 2 dose levels of panobinostat will be tested. Up to 6participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of panobinostat is found.

All participants will receive the same dose level of ICE.

Once the highest tolerable dose is found, up to 20 extra participants, called the expansion group, will receive the study drugs at that dose.

Study Drug Administration:

Each cycle is 14 days.

ICE Administration:

On Day 1 (+/- 2 days) of Cycles 1-3, you will receive ifosfamide by vein over 24 hours.

On Day 1 (+/- 2 days) of Cycles 1-3, you will receive carboplatin by vein over 1 hour.

On Days 1-3 (+/- 2 days) of Cycles 1-3, you will receive etoposide by vein over 2 hours.

You will also receive mesna to help prevent side effects. On Day 2 (+/- 2 days) of Cycles 1-3, you will receive mesna by vein over 12 hours.

You will also receive pegfilgrastim to help prevent side effects. Beginning 24-48 hours after the completion of chemotherapy of Cycles 1-3, you will take pegfilgrastim through a needle under the skin.

Panobinostat Administration:

You will take panobinostat by mouth starting Day -6 of Cycle 1 (6 days before your first dose of ICE). You will take the panobinostat on Days -6, -4, and -2 of Cycle 1 and Days 1, 3, 5, 8, 10, and 12 of Cycles 1 and 2.

If you are in the expansion group, you will take panobinostat by mouth starting Day -6 of Cycle 1 (6 days before your first dose of ICE). You will take the panobinostat on Days -6, -4, and -2 of Cycle 1 and Days 1, 3, and 5 of Cycles 1 and 2.

You should take panobinostat around the same time each day with 1 cup (8 ounces) of water. You should swallow the capsules whole and not chew them. You must avoid grapefruit or grapefruit juice and seville (sour) oranges while on study.

If you miss a dose of panobinostat, take it as soon as you remember it on the same day. However, if more than 12 hours have passed since you were supposed to take the dose, you should skip that day's dose. In that case, wait to take panobinostat until the next scheduled dosing day.

Study Visits:

On Days -6 and -2 of Cycle 1, you will have 2 ECGs.

Within 7 days before each ICE therapy:

* You will have a physical exam, including measurement of your height, weight, and vital signs.
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* You will be asked if you have had any side effects.

One (1) time a week, blood (2 1/2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond, you will have an ECG.

After Cycle 3:

* You will have a CT scan of your head and neck, chest, abdomen, and pelvis to check the status of the disease.
* If your bone marrow was positive at screening, you will have a positron emission tomography (PET) scan to check the status of the disease.

Length of Study:

You be on study for up to 3 cycles (about 42 days). You will be taken off study early if the disease worsens or you experience intolerable side effects.

End-of-Study Visit:

After you are off study, you will have an end-of-study visit at which the following will be performed:

You will have a physical exam, including measurement of your weight and vital signs.

You will have an ECG.

This is an investigational study. Panobinostat is not FDA approved or commercially available. It is currently being used for research purposes only.

ICE is FDA approved and commercially available for the treatment of several types of lymphoma, including relapsed and refractory Hodgkins lymphoma. The combination of panobinostat and ICE for the treatment of Hodgkin's lymphoma is investigational.

Up to 102 patients will take part in this study. All will be enrolled at MD Anderson.

Phase II:

The Study Drugs:

Panobinostat is designed to block the function of enzymes that are found inside cancer cells. These enzymes trigger cells to grow and multiply out of control. By blocking these enzymes, it may slow down the growth of or kill cancer cells.

Ifosfamide is designed to slow or stop the growth of cancer cells.

Carboplatin is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

Etoposide is designed to block cell growth.

Baseline Tests:

If you are found to be eligible to take part in this study, the following tests and procedures will be performed about 7 days before the first dose of the study drug:

* You will have a physical exam, including measurement of your height, weight, and vital signs (blood pressure and heart rate).
* You will have 1 electrocardiogram (ECG -- a test that measures the electrical activity of the heart).
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* Women who are able to become pregnant must have a negative blood (about 1 1/2 teaspoons) pregnancy test.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups.

* If you are in Group 1, you will receive ICE.
* If you are in Group 2, you will receive ICE and panobinostat.

Study Drug Administration:

Each cycle is 14 days.

ICE Administration:

On Day 1 (+/- 2 days) of Cycles 1-3, you will receive ifosfamide by vein over 24 hours.

On Day 1 (+/- 2 days) of Cycles 1-3, you will receive carboplatin by vein over 1 hour.

On Days 1-3 (+/- 2 days) of Cycles 1-3, you will receive etoposide by vein over 2 hours.

You will also receive mesna to help prevent side effects. On Day 2 (+/- 2 days) of Cycles 1-3, you will receive mesna by vein over 12 hours.

You will also receive pegfilgrastim to help prevent side effects. Beginning 24-48 hours after the completion of chemotherapy of Cycles 1-3, you will take pegfilgrastim through a needle under the skin.

Panobinostat Administration:

If you are in a group that will receive panobinostat, you will take panobinostat by mouth starting Day -6 of Cycle 1 (6 days before your first dose of ICE). You will take the panobinostat on 3 times a week during Cycles 1 and 2 (Days -6, -4, and -2 of Cycle 1 and Days 1, 3, and 5 Cycles 1 and 2).

You should take panobinostat around the same time each day with 1 cup (8 ounces) of water. You should swallow the capsules whole and not chew them. You must avoid grapefruit or grapefruit juice and seville (sour) oranges while on study.

If you miss a dose of panobinostat, take it as soon as you remember it on the same day. However, if more than 12 hours have passed since you were supposed to take the dose, you should skip that day's dose. In that case, wait to take panobinostat until the next scheduled dosing day.

Study Visits:

On Days -6 and -2 of Cycle 1, you will have 2 ECGs.

Within 7 days before each ICE therapy:

* You will have a physical exam, including measurement of your height, weight, and vital signs.
* Blood (about 2 1/2 teaspoons) will be drawn for routine tests.
* You will be asked if you have had any side effects.

One (1) time a week, blood (2 1/2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and beyond, you will have an ECG.

After Cycle 3:

* You will have a CT scan of your head and neck, chest, abdomen, and pelvis to check the status of the disease.
* If your bone marrow was positive at screening, you will have a PET scan to check the status of the disease.

Length of Study:

You be on study for up to 3 cycles (about 42 days). You will be taken off study early if the disease worsens or you experience intolerable side effects.

End-of-Study Visit:

After you are off study, you will have an end-of-study visit at which the following will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will have an ECG.

This is an investigational study. Panobinostat is not FDA approved or commercially available. It is currently being used for research purposes only.

ICE is FDA approved and commercially available for the treatment of several types of lymphoma, including relapsed and refractory Hodgkins lymphoma. The combination of panobinostat and ICE for the treatment of Hodgkin's lymphoma is investigational.

Up to 102 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed classical Hodgkin lymphoma (nodular sclerosis, mixed cellularity, or lymphocyte-rich classical HL).
2. Patients must have failed (relapsed or refractory) front-line standard anthracycline-containing regimen, such as ABVD, Stanford V, or BEACOPP.
3. Bidimensionally measurable disease with at least 1 lesion >/= 2.0 cm in a single dimension
4. Acceptable hematologic status:Hemoglobin >/= 9.0 g/dL, Absolute neutrophil count >/= 1500 cells/mm3, Platelet count >/= 100,000 cells/mm3
5. Normal serum K+, Mg+, PO4, and total Ca++ (pre-treatment abnormal values may be therapeutically corrected before starting therapy and must be documented as normal or if abnormal values persist must be documented as clinically insignificant). Albumin should be >/= 3
6. Pre-study World Health Organization (WHO) performance status of 0, 1, or 2
7. Age >/= 16 years
8. Voluntary signed Institutional Review Board (IRB) approved consent informed before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
9. Patients of reproductive potential (female of child bearing potential has not been postmenopausal for at least 12 consecutive months or not surgically sterile; male of child bearing potential has not been surgically sterile)must follow accepted birth control methods (e.g. barrier method) during treatment.
10. Clinically euthyroid. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
11. Baseline Multiple Gated Acquisition (MUGA) or ECHO must demonstrate left ventricular ejection fraction (LVEF) >/= 50%.

Exclusion Criteria:

1. Lymphocyte predominant histology
2. More than one prior chemotherapy regimens.
3. Prior therapy with other HDAC inhibitors, including valproic acid
4. Prior therapy with heat shock protein (HSP)-90 inhibitors
5. Prior stem cell transplant
6. Abnormal liver function: Bilirubin > 2.0 mg/dL (26 µmol/L), Alkaline phosphatase > 2 x upper limits of normal (ULN), aspartate aminotransferase AST (SGOT) and/or alanine aminotransferase ALT > 2 x ULN
7. Serum creatinine >1.5 mg/dl
8. Presence of Central Nervous System (CNS) involvement with Hodgkin lymphoma
9. Presence of Human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS).
10. Another primary malignancy (other than squamous cell and basal cell carcinoma of the skin, in situ carcinoma of the cervix, or treated prostate cancer with a stable Prostate Specific Antigen PSA) for which the patient has not been disease free for at least 3 years.
11. Serious nonmalignant disease (e.g., congestive heart failure, hydronephrosis); active uncontrolled bacterial, viral, or fungal infections; or other conditions which would compromise protocol objectives in the opinion of the investigator
12. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:History or presence of sustained ventricular tachyarrhythmia, Any history of ventricular fibrillation or torsade de pointes, Bradycardia defined as HR< 50 bpm, Patients with pacemakers are eligible if HR >/= 50 bpm, Screening ECG with a corrected QT interval (QTc) > 450 msec, Right bundle branch block + left anterior hemiblock (bifascicular block), Patients with myocardial infarction or unstable angina </= 6 months prior to starting study drug, Other clinically significant heart disease (e.g., congestive heart failure (CHF) New York Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
13. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum Beta-human chorionic gonadotropin (Beta-hCG) pregnancy test result obtained during screening, unless the female has recently (within 8 weeks) undergone egg harvest, which would result in the (Beta-hCG) test to be elevated without pregnancy. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
14. Patient has received other investigational drugs within 14 days before enrollment or who have not recovered from side effects of those therapies.
15. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
16. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat
17. Patients with diarrhea > Common Terminology Criteria for Adverse Events Version 4 (CTCAE V.4) grade 2
18. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug.
19. Patients who have received either immunotherapy within </= 8 weeks; chemotherapy within </= 3 weeks; or radiation therapy to > 30% of marrow-bearing bone within </= 2 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
20. Patients who have undergone major surgery </= 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-01-31 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiro Oki, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 2011 to March 2016
Pre-assignment Details: 62 participants enrolled, 3 participants not treated on the study (1) adverse event (1) financial issue, and (1) consent withdrawal.
Groups:
- Phase I: Panobinostat + ICE 10 mg; Phase I: Panobinostat + ICE 20 mg; Phase I: Panobinostat + ICE 30 mg: The dose level for ICE is fixed. Patients received Panobinostat daily on Mon-Wed-Fri starting one week prior to cycle 1of ICE and during two weeks of C1-2 of ICE. Pre-defined dose levels of Panobinostat: Dose level -1 = 10 mg Dose level 0 = 20 mg: Dose level 1= 30 mg
- Phase II: Standard of Care (ICE); Phase II: Panobinostat + ICE: Patients are randomized between ICE and Panobinostat plus ICE arms using A Bayesian adaptive algorithm. The dose level for Panobinostat was determined to be dose level 1 at 30mg as MTD during the phase I expansion cohort.
Period: Overall Study
Arm/Group | Phase I: Panobinostat + ICE 10 mg | Phase I: Panobinostat + ICE 20 mg | Phase I: Panobinostat + ICE 30 mg | Phase II: Standard of Care (ICE) | Phase II: Panobinostat + ICE
Started | 3 | 6 | 20 | 13 | 14
Completed | 3 | 6 | 17 | 12 | 11
Not Completed | 0 | 0 | 3 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Screen failure | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Panobinostat + ICE 10 mg | Phase I: Panobinostat + ICE 20 mg | Phase I: Panobinostat + ICE 30 mg | Phase II: Standard of Care (ICE) | Phase II: Panobinostat + ICE | Total
Number analyzed (Participants) | 3 | 6 | 20 | 12 | 11 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 19 | 12 | 10 | 50
  >=65 years | 0 | 0 | 1 | 0 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 9 | 9 | 7 | 28
  Male | 2 | 4 | 11 | 3 | 4 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 5 | 1 | 1 | 8
  White | 3 | 5 | 15 | 11 | 10 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 20 | 12 | 11 | 52

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Panobinostat + ICE
Description: Maximum Tolerated Dose (MTD) of Panobinostat + ICE
Time Frame: From first dose of panobinostat (or chemotherapy, in the arm of ICE alone) until 30 days after last dose, up to 6 years
Measure: Number; unit: mg
Groups:
- Phase I: Panobinostat + ICE (Maximal Tolerated Dose (MTD): The dose level for ICE is fixed. Patients received Panobinostat daily on Mon-Wed-Fri starting one week prior to cycle 1of ICE and during two weeks of C1-2 of ICE. Pre-defined dose levels of Panobinostat: Dose level -1 = 10 mg Dose level 0 = 20 mg: Dose level 1= 30 mg
Arm/Group | Phase I: Panobinostat + ICE (Maximal Tolerated Dose (MTD)
Number analyzed (Participants) | 29
mg | 30

2. Primary Outcome: Number of Participants With Complete Remission (CR)
Description: Will be assessed by Kaplan-Meier methods.
Time Frame: Assessed after 3 cycles of ICE (2 months)
Population: Per protocol all Phase I Cohorts are analyzed as a single group.
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Panobinostat + ICE: Patients are randomized between ICE and Panobinostat plus ICE arms using A Bayesian adaptive algorithm. The dose level for Panobinostat was determined to be dose level 1 at 30mg as MTD during the phase I expansion cohort.
Arm/Group | Phase I: Panobinostat + ICE (Maximal Tolerated Dose (MTD) | Phase II: Standard of Care (ICE) | Phase II Panobinostat + ICE
Number analyzed (Participants) | 29 | 12 | 11
Participants
  Complete Response | 21 | 8 | 9
  Partial Response | 4 | 1 | 0
  Stable Disease | 2 | 2 | 2
  Progressive Disease | 2 | 1 | 0

3. Secondary Outcome: Percentage of Participants With Failure Free Survival (FFS)
Description: FFS duration was calculated from date of study entry to date of progression or death or change of therapy, whichever came first.
Time Frame: 16 months
Population: Per protocol all Phase I Cohorts are analyzed as a single group.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I: Panobinostat + ICE (Maximal Tolerated Dose (MTD) | Phase II: Standard of Care (ICE) | Phase II Panobinostat + ICE
Number analyzed (Participants) | 29 | 12 | 11
percentage of participants | 61 | 82 | 75

ADVERSE EVENTS:
Time Frame: All AE were recorded from first dose of panobinostat (or chemotherapy, in the arm of ICE alone) until 30 days after last dose.
Groups:
- Phase I: Panobinostat + ICE 10 mg; Phase I: Panobinostat + ICE 20 mg; Phase I: Panobinostat + ICE 30 mg: The dose level for ICE is fixed. Patients received Panobinostat daily on Mon-Wed-Fri starting one week prior to cycle 1 of ICE and during two weeks of C 1-2 of ICE. Pre-defined dose levels of Panobinostat: Dose level -1 = 10 mg Dose level 0 = 20 mg: Dose level 1= 30 mg
- Phase II: Panobinostat+ICE: Participants are randomized between ICE and Panobinostat plus ICE arms using A Bayesian adaptive algorithm. The dose level for Panobinostat was determined to be dose level 1 at 30mg as MTD during the phase I expansion cohort.
Arm/Group | Phase I: Panobinostat + ICE 10 mg | Phase I: Panobinostat + ICE 20 mg | Phase I: Panobinostat + ICE 30 mg | Phase II: Standard of Care (ICE) | Phase II: Panobinostat+ICE
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/20 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 20/20 | 12/12 | 11/11
Other Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 19/20 | 12/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Panobinostat + ICE 10 mg (N=3) | Phase I: Panobinostat + ICE 20 mg (N=6) | Phase I: Panobinostat + ICE 30 mg (N=20) | Phase II: Standard of Care (ICE) (N=12) | Phase II: Panobinostat+ICE (N=11)
Neutropenia (Investigations) | 0 | 0 | 11 | 3 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 11 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 19 | 9 | 11
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 11 | 6 | 11
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0
Syncope (Cardiac disorders) | 0 | 0 | 1 | 3 | 0
Dizziness (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (Cardiac disorders) | 0 | 0 | 0 | 3 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Panobinostat + ICE 10 mg (N=3) | Phase I: Panobinostat + ICE 20 mg (N=6) | Phase I: Panobinostat + ICE 30 mg (N=20) | Phase II: Standard of Care (ICE) (N=12) | Phase II: Panobinostat+ICE (N=11)
Nausea (Gastrointestinal disorders) | 0 | 1 | 19 | 12 | 9
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 11 | 9 | 7
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 10 | 3 | 7
Mucositis (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 5
Neutropenia (Investigations) | 0 | 0 | 19 | 5 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 12 | 1 | 1
Thrombocytopenia (Investigations) | 0 | 1 | 19 | 11 | 11
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 19 | 10 | 11
AST (Investigations) | 0 | 1 | 4 | 1 | 2
ALT (Investigations) | 0 | 1 | 6 | 1 | 2
Hyperbilirubinemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 4 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 7 | 5 | 4
Syncope (Cardiac disorders) | 0 | 0 | 1 | 3 | 0
Dizziness (Cardiac disorders) | 0 | 0 | 5 | 1 | 2
Fatigue (Cardiac disorders) | 0 | 1 | 18 | 12 | 10
Dehydration (Cardiac disorders) | 0 | 0 | 1 | 2 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT01169636/Prot_SAP_000.pdf